CLINICAL TRIAL: NCT00110409
Title: Trial of Asthma Patient Education in the Emergency Room
Brief Title: Asthma Patient Education in the Emergency Room
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital for Special Surgery, New York (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Carol A. Mancuso, MD, Hospital for Special Surgery
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 173; R01HL075893 (NIH)
Record Dates: First submitted 2005-05-06; First posted 2005-05-09 (Estimated); Last update posted 2013-06-10 (Estimated); Status verified 2013-06

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Intervention participants will receive information focusing on asthma self-management, education, self-efficacy, and social support while in the hospital emergency room. Telephone reinforcement will occur for 8 weeks following study entry.
  Interventions: Behavioral: Asthma Education in Adults
- 2 (Active Comparator): Participants in the control group will receive standard emergency room education about asthma.
  Interventions: Behavioral: Standard Emergency Room Asthma Education

INTERVENTIONS:
Behavioral: Asthma Education in Adults — The intervention involves enhancing asthma education, asthma self-efficacy and asthma-related social support and is administered during a single in-person session in the ED (or hospital for admitted patients) followed by telephone reinforcement.
  Arms: 1
Behavioral: Standard Emergency Room Asthma Education — Participants will receive standard emergency room education about asthma.
  Arms: 2

SUMMARY:
The objective of this randomized trial is to assess the effectiveness of an intervention involving education, self-efficacy, and social support in improving quality of life outcomes among 296 adult asthma patients treated in the emergency room. The main outcome will be a comparison of within-patient change in quality of life between enrollment and 8 weeks. Secondary objectives will be to assess the effectiveness of the intervention in decreasing the need for rescue inhaled beta agonists, in improving peak flow meter rates, and in decreasing the number of days lost from work or school due to asthma. These outcomes will be measured again at 16 weeks to determine if benefits are sustained. Additional outcomes at 16 weeks and 1 year will be to assess the effectiveness of the intervention in decreasing urgent resource utilization for asthma and cost effectiveness.

DETAILED DESCRIPTION:
BACKGROUND:

Many urban asthma emergency room patients lack effective self-management. Most current training programs are administered in outpatient settings and have low attendance rates for emergency room patients. There is a great need to develop effective programs that can be easily administered in the emergency room for patients who, in many cases, are not present in other settings to receive education. This proposal builds on preliminary studies and is tailored to provide emergency room patients with basic education during "a teachable moment" when they may be most receptive to asthma information.

DESIGN NARRATIVE:

Patients will be recruited from two New York City urban emergency rooms or inpatient settings and randomized to the intervention or control groups. Intervention patients will receive a protocol focusing on asthma self-management, education, self-efficacy, and social support, with telephone reinforcement for 8 weeks. Control patients will receive standard emergency room education about asthma.

ELIGIBILITY:
Inclusion Criteria:

* Patients will be eligible if they are 18 years of age or older
* Fluent in English
* Have a known diagnosis of asthma
* Will receive treatment for asthma during the current hospitalization or emergency room visit.

Exclusion Criteria:

* Cognitive deficits
* Other pulmonary diseases or severe comorbidity
* Do not have out-patient access to a telephone

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 296 (Estimated)
Dates: Start 2005-01; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Quality of life | Measured at 8 weeks

SECONDARY OUTCOMES:
Rescue inhaled beta agonist use | Measured at 8 weeks
Peak flow meter rates | Measured at 8 weeks
Number of days lost from work or school due to asthma | Measured at 8 weeks
Decreasing urgent resource utilization for asthma | Measured at 16 weeks and 1 year
Cost effectiveness | Measured at 16 weeks and 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Carol A. Mancuso, MD, Study Chair — Hospital for Special Surgery, New York
Locations (1):
- New York, New York, United States

REFERENCES:
- [Background] Mancuso CA, Peterson MG. Different methods to assess quality of life from multiple follow-ups in a longitudinal asthma study. J Clin Epidemiol. 2004 Jan;57(1):45-54. doi: 10.1016/S0895-4356(03)00248-8. PMID 15019010
- [Background] Mancuso CA, Rincon M, Robbins L, Charlson ME. Patients' expectations of asthma treatment. J Asthma. 2003 Dec;40(8):873-81. doi: 10.1081/jas-120023578. PMID 14736086
- [Background] Mancuso CA, Rincon M, Charlson ME. Adverse work outcomes and events attributed to asthma. Am J Ind Med. 2003 Sep;44(3):236-45. doi: 10.1002/ajim.10257. PMID 12929143
- [Background] Mancuso CA, Rincon M, McCulloch CE, Charlson ME. Self-efficacy, depressive symptoms, and patients' expectations predict outcomes in asthma. Med Care. 2001 Dec;39(12):1326-38. doi: 10.1097/00005650-200112000-00008. PMID 11717574
- [Background] Mancuso CA, Peterson MG, Charlson ME. Effects of depressive symptoms on health-related quality of life in asthma patients. J Gen Intern Med. 2000 May;15(5):301-10. doi: 10.1046/j.1525-1497.2000.07006.x. PMID 10840265
- [Derived] Peterson MG, Gaeta TJ, Birkhahn RH, Fernandez JL, Mancuso CA. History of symptom triggers in patients presenting to the emergency department for asthma. J Asthma. 2012 Aug;49(6):629-36. doi: 10.3109/02770903.2012.690480. Epub 2012 Jun 28. PMID 22742414